CLINICAL TRIAL: NCT01789255
Title: A Pilot Trial of Vorinostat Plus Tacrolimus and Methotrexate to Prevent Graft Versus Host Disease Following Unrelated Donor Hematopoietic Stem Cell Transplantation
Brief Title: Vorinostat, Tacrolimus, and Methotrexate in Preventing GVHD After Stem Cell Transplant in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NCI-2013-00355; NCI-2013-00355 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00070080; UMCC 2012.047 (Other: University of Michigan University Hospital); 9330 (Other: CTEP); P30CA046592 (NIH)
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; B-cell Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Graft Versus Host Disease; Intraocular Lymphoma; Myelodysplastic Syndrome With Isolated Del(5q); Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Post-transplant Lymphoproliferative Disorder; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Ringed Sideroblasts; Refractory Chronic Lymphocytic Leukemia; Refractory Cytopenia With Multilineage Dysplasia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Central Nervous System Hodgkin Lymphoma; Secondary Central Nervous System Non-Hodgkin Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Graft vs Host Disease; Intraocular Lymphoma; Chromosome 5q Deletion Syndrome; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia | interventions — Vorinostat; Tacrolimus; Cyclosporine; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (vorinostat, tacrolimus, methotrexate) (Experimental): Patients receive vorinostat PO BID on days -10 to 100. Beginning on day -3, patients receive tacrolimus IV continuously or PO BID (or cyclosporine IV continuously or PO in patients unable to tolerate tacrolimus) with taper on days 100-180.Patients also receive methotrexate IV QD on days 1, 3, 6, and 11.
  Interventions: Drug: vorinostat; Drug: tacrolimus; Drug: cyclosporine; Drug: methotrexate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This pilot phase II trial studies how well giving vorinostat, tacrolimus, and methotrexate works in preventing graft-versus-host disease (GVHD) after stem cell transplant in patients with hematological malignancies. Vorinostat, tacrolimus, and methotrexate may be an effective treatment for GVHD caused by a bone marrow transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and the feasibility of the addition of vorinostat to tacrolimus and methotrexate GVHD prophylaxis.

SECONDARY OBJECTIVES:

I. To determine day 100 grades 2-4 acute GVHD. II. To determine 1-year overall survival and relapse-free survival. III. To correlate plasma concentrations of inflammatory markers of acute GVHD. IV. To correlate protein acetylation in peripheral blood mononuclear cells before and after administration of vorinostat.

OUTLINE:

Patients receive vorinostat orally (PO) twice daily (BID) on days -10 to 100. Beginning on day -3, patients receive tacrolimus intravenously (IV) continuously or PO BID (or cyclosporine IV continuously or PO in patients unable to tolerate tacrolimus) with taper on days 100-180.Patients also receive methotrexate IV once daily (QD) on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed up periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* A prospective patient for allogeneic HSCT for hematologic conditions, both malignant and non-malignant; donor can be unrelated marrow or peripheral blood cells; a patient with history of central nervous system (CNS) involvement is eligible if CNS disease is in remission at time of study consideration
* The donor and recipient must have a human leukocyte antigen (HLA)-8/8 allelic match at the HLA-A, -B, -C, and -DRB1; high-resolution typing is required for all alleles
* Diagnoses to be included:
* Acute myelogenous leukemia at the following stages:

  * First remission
  * Second or subsequent remission
  * Complete remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment and < 5% blasts in the bone marrow
* Chronic myelogenous leukemia at the following stages:

  * First or subsequent chronic phase:

    * Patient refused tyrosine kinase therapy or is otherwise not suited for it
    * Stable, not hematologic remission: blasts present in marrow and/or peripheral blood, but disease does not qualify as accelerated or blast phase
    * Hematologic remission: no blast cells or precursor cells in the blood or marrow
    * Partial cytogenetic remission: Philadelphia chromosome positive (Ph+) metaphases > 0% but < 35%
    * Complete cytogenetic remission: absence of Ph+ metaphases
  * Accelerated phase - any one of the following symptoms:

    * White blood cells (WBC) difficult to control (> 50 x 10^9/L despite therapy)
    * Rapid doubling of WBC (< 5 days)
    * 10% blasts in blood or marrow
    * 20% blasts and/or promyelocytes in blood or marrow
    * 20% basophils and/or eosinophils in blood
    * Anemia or thrombocytopenia unresponsive to standard treatment
    * Persistent thrombocytosis (> 1000 x 10^9/L)
    * Cytogenetic abnormalities in addition to Ph+
    * Increasing splenomegaly
    * Marrow fibrosis
* Myelodysplastic syndromes at any of the following stages:

  * Refractory anemia
  * Refractory anemia with ringed sideroblasts
  * Refractory cytopenia with multilineage dysplasia
  * Refractory cytopenia with multilineage dysplasia and ringed sideroblasts
  * Refractory anemia with excess blasts-1 (5-10% blasts)
  * Refractory anemia with excess blasts-2 (10-20% blasts)
  * Myelodysplastic syndrome, unclassified
  * Myelodysplastic syndrome (MDS) associated with isolated del (5q)
  * Chronic myelomonocytic leukemia
* Primary Myelofibrosis

  * Intermediate-2 risk or high risk disease
  * Patients should have extinguished standard of care options prior to being considered for this trial
* Chronic lymphocytic leukemia

  * Complete remission: the disease is completely absent and no relapse occurred prior to the preparative regimen; requires all of the following:

    * Nodular partial remission: complete response with persistent lymphoid nodules in bone marrow
    * Partial remission: reduction of more than 50% in the disease burden regardless of the number of lines of therapy received
* Mature B cell malignancies

  * Patients should have extinguished standard of care options prior to being considered eligible for this trial
  * First complete remission (CR1) confirmed: complete disappearance of all known disease; the term "confirmed" is defined as a laboratory and/or pathological or radiographic determination.
  * CR1 unconfirmed (CRU1): complete disappearance of all known disease with the exception of persistent scan abnormalities of unknown significance; the term "unconfirmed" is defined as scan abnormalities of unknown significance that are not biopsied or otherwise evaluated
  * Second or subsequent complete remission (CR2+) confirmed: the recipient relapsed, then achieved complete absence of disease without radiographic evidence of disease
  * CR2+ unconfirmed: the recipient has achieved a second or subsequent complete response but has persistent radiographic abnormalities of unknown significance.
  * Partial remission: reductions of >= 50% in greatest diameter of all sites of known disease and no new sites
* Karnofsky >= 70%
* Life expectancy of greater than 6 months
* Total bilirubin =< 2.5 mg% (unless from Gilbert's disease or disease-related)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3.0 X institutional upper limit of normal
* Estimated or actual glomerular filtration rate (GFR) > 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal; GFR should be corrected for body surface area (BSA)
* Diffusing capacity of the lung for carbon monoxide (DLCO) > 50%; DLCO should be corrected for hemoglobin
* Forced expiratory volume in 1 second (FEV1) > 50%
* Forced vital capacity (FVC) > 50%
* Ejection fraction >= 50%
* The effects of vorinostat on the developing human fetus are unknown; for this reason and because histone deacetylase inhibitor agents as well as other therapeutic agents used in this trial (e.g., tacrolimus and methotrexate) are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of vorinostat administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients must be able to swallow capsules/tablets

Exclusion Criteria:

* Patients who are not a candidate for an unrelated donor allogeneic HSCT based on the current institutional bone marrow transplant (BMT) program clinical practice guidelines; organ function criteria will be utilized per the current institutional BMT program clinical practice guidelines; there will be no restriction to study entry based on hematological parameters
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* Patients undergoing a total body irradiation (TBI)-based conditioning regimen (TBI 1200 centigray [cGy])
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients still under therapy for presumed or proven infection are eligible provided there is clear evidence (radiographic findings and/or culture results) that the infection is well-controlled; patients under treatment for infection will be enrolled only after clearance from the Principal Investigator (PI)
* Pregnant women are excluded from this study because vorinostat is a histone deacetylase inhibitor agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated with vorinostat
* Patients with evidence of human immunodeficiency virus (HIV) seropositivity and/or positive polymerase chain reaction (PCR) assay, human T-lymphotropic virus (HTLV)1/HTLV2 seropositivity; the safety of allogeneic HSCT is not yet well-established for this population
* Patients with evidence of hepatitis B or hepatitis C PCR positivity; hepatitis reactivation following myelosuppressive therapy can lead to fatal complications
* Patients with a history of prolonged corrected QT interval (QTc) syndrome
* Patients asking or who have had prior treatment with a drug like vorinostat (i.e., valproic acid) within the last 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Reddy, Principal Investigator — University of Michigan University Hospital
Locations (1):
- University of Michigan University Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care (Vorinostat, Tacrolimus, Methotrexate): Patients receive vorinostat PO BID on days -10 to 100. Beginning on day -3, patients receive tacrolimus IV continuously or PO BID (or cyclosporine IV continuously or PO in patients unable to tolerate tacrolimus) with taper on days 100-180. Patients also receive methotrexate IV QD on days 1, 3, 6, and 11.
Period: Overall Study
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [45 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants That Experience Grade 2-4 Acute GVHD (Graft Versus Host Disease) by Day 100
Description: The incidence of grade 2-4 acute GVHD (Graft Versus Host Disease) by day 100
  Grade 2 GVHD: Maculopapular rash covering 25-50% of BSA (Body Surface Area), bilirubin between 3.1-6 mg/dl, and/ or adult stool output between 1000-1500 ml/day (child between 20-30 ml/kg/day).
  Grade 3 GVHD: Maculopapular rash covering >50% of BSA, bilirubin between 6.1-15 mg/dl, and/ or adult stool output >1500 ml/day (child >30 ml/kg/day).
  Grade 4 GVHD: Generalized erythroderma plus bullous formation and desquamation >5% BSA, bilirubin >15 mg/dl, and/ or severe abdominal pain with or without ileus, or grossly bloody stool.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 12
participants | 2

2. Secondary Outcome: Mean Percent of Planned Dose Administered
Description: The addition of vorinostat to tacrolimus and methotrexate for GVHD prophylaxis will be considered feasible if 60% or more of the planned doses are administered.
Time Frame: Up to day 30
Measure: Mean (Full Range); unit: percent of dose administered
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 12
percent of dose administered | 82.5 [53.8 to 100]

3. Secondary Outcome: The Percentage of Patients Alive Without GVHD or Use of Steroids
Description: The percentage of patients alive without GVHD or use of steroids at 1 year.
Time Frame: Up to 1 year
Population: This trial consisted of an initial pilot phase, funded by the NCI, that enrolled 12 patients (NCT01789255). The trial was extended to enroll an additional 25 patients. The results presented here include information for all 37 patients. The analysis population description for all 37 patients can be found under NCT01790568.
Measure: Number; unit: percentage of patients
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 37
percentage of patients | 47

4. Secondary Outcome: The Percentage of Patients Alive at 1 Year
Description: The percentage of patients alive at 1 year
Time Frame: Up to 1 year
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 37
percentage of patients | 76

5. Secondary Outcome: The Percentage of Patients With Relapse at 1 Year
Time Frame: Up to 1 year
Measure: Number; unit: percentage of patients
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 12
percentage of patients | 19

6. Secondary Outcome: Median Ac-H3 Levels in Patients Treated With Vorinostat and Patients Not Treated With Vorinostat
Description: Median Ac-H3 levels ( depicted as a ratio of ac-H2 optical density (OD) and beta actin OD) were compared in patients treated with Vorinostat to patients not treated with Vorinostat. Optical Density is a dimensionless unit.
Time Frame: Up to day 100
Population: as for outcome 3
Measure: Median (Full Range); unit: Ratio
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 37
Ratio
  Treated with Vorinostat | 0.943 [0.42 to 1.27]
  Not Treated with Vorinostat | 0.679 [0.19 to 1.01]
Statistical Analysis 1: Comparison: Supportive Care (Vorinostat, Tacrolimus, Methotrexate); Test type: Other; p = 0.02642, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Median Plasma Concentration of IL-6 in Patients Treated With Vorinostat and Patients Not Treated With Vorinostat
Description: Median plasma concentration of IL-6 (Interleukin-6 cytokine) was compared in patients treated with Vorinostat to those not treated with Vorinostat.
Time Frame: Up to day 100
Population: as for outcome 3
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Number analyzed (Participants) | 37
pg/mL
  Treated with Vorinostat | 4.2 [0.1 to 22.3]
  Not Treated with Vorinostat | 7.6 [0.3 to 70.1]
Statistical Analysis 1: Comparison: Supportive Care (Vorinostat, Tacrolimus, Methotrexate); Test type: Other; p = 0.028, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Supportive Care (Vorinostat, Tacrolimus, Methotrexate)
Serious Adverse Events (participants affected / at risk) | 7/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Vorinostat, Tacrolimus, Methotrexate) (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Immune system disorders, Other (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified, Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Vorinostat, Tacrolimus, Methotrexate) (N=12)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Immune system disorders, Other (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 8 (8)
White blood cell decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified, Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less